CLINICAL TRIAL: NCT00001395
Title: Long Term Follow-Up of Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940106; 94-EI-0106
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-03

CONDITIONS: Blindness; Cataract; Diabetes Mellitus; Diabetic Retinopathy; Macular Degeneration
Keywords: Cataracts; Complications; Rates of Progression; Diabetic Retinopathy
MeSH Terms: conditions — Blindness; Cataract; Diabetes Mellitus; Diabetic Retinopathy; Macular Degeneration

SUMMARY:
The efficacy of laser photocoagulation treatment for diabetic retinopathy has been demonstrated by several National Eye Institute (NEI) sponsored clinical trials. The Diabetic Retinopathy Study (DRS) demonstrated that scatter photocoagulation reduces the risk of blindness from diabetic retinopathy. The Early Treatment Diabetic Retinopathy Study (ETDRS) extended these findings by providing information on when to initiate scatter photocoagulation and by demonstrating that focal treatment was effective in treating macula edema. The Krypton Argon Regression Neovascularization Study (KARNS) showed that scatter photocoagulation with krypton red laser was just as safe and effective as the argon blue-green laser in the treatment of proliferative diabetic retinopathy.

Unfortunately, there is little data on the long term effects of photocoagulation on visual function. The first objective of this study is to assess the long term effects of photocoagulation for diabetic retinopathy. A second objective is to provide additional information on the risk of progression of cataracts in persons with diabetes. All patients previously treated with laser photocoagulation (focal and/or scatter) are eligible to participate in this long term study. The first priority will be given to patients who participated in the ETDRS and KARNS because of the wealth of information available regarding the details of their treatment and course after treatment. Study evaluations will include a standard ophthalmic examination, fluorescein angiography, lens and fundus photography.

DETAILED DESCRIPTION:
The efficacy of laser photocoagulation treatment for diabetic retinopathy has been demonstrated by several National Eye Institute (NEI) sponsored clinical trials. The Diabetic Retinopathy Study (DRS) demonstrated that scatter photocoagulation reduces the risk of blindness from diabetic retinopathy. The Early Treatment Diabetic Retinopathy Study (ETDRS) extended these findings by providing information on when to initiate scatter photocoagulation and by demonstrating that focal treatment was effective in treating macula edema. The Krypton Argon Regression Neovascularization Study (KARNS) showed that scatter photocoagulation with krypton red laser was just as safe and effective as the argon blue-green laser in the treatment of proliferative diabetic retinopathy.

Unfortunately, there is little data on the long term effects of photocoagulation on visual function. The first objective of this study is to assess the long term effects of photocoagulation for diabetic retinopathy. A second objective is to provide additional information on the risk of progression of cataracts in persons with diabetes. All patients previously treated with laser photocoagulation (focal and/or scatter) are eligible to participate in this long term study. The first priority will be given to patients who participated in the ETDRS and KARNS because of the wealth of information available regarding the details of their treatment and course after treatment. Study evaluations will include a standard ophthalmic examination, fluorescein angiography, lens and fundus photography.

ELIGIBILITY:
All patients with diabetic retinopathy that has been treated previously with laser photocoagulation, either focal or scatter treatment, are eligible.

Patients must be 18 or more years of age.

Patients who have not had laser photocoagulation for diabetic retinopathy are not eligible for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 1994-03; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States